CLINICAL TRIAL: NCT04493892
Title: Hair Care Product Use Among Women Of Color: A Northern Manhattan Intervention
Brief Title: Hair Care Product Use Among Women Of Color
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Jasmine McDonald, Assistant Professor of Epidemiology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAS9968; 5P30ES009089 (NIH)
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer; Pregnancy Related; Exposure During Pregnancy
Keywords: Hair products; Phthalates; Endocrine disrupting chemicals
MeSH Terms: conditions — Breast Neoplasms | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Intervention (Experimental): All participants receive educational information on the potential health risk of endocrine disruptor chemicals in hair care products, specifically phthalates. Provide information on how to reduce exposure.
  Interventions: Behavioral: Educational Intervention

INTERVENTIONS:
Behavioral: Educational Intervention — Deliver an educational intervention on harmful chemical exposures, such as phthalates, found in hair care products, developed by the research team using empirical evidence with key informant feedback. The intervention will cover phthalates 1) Exposure through HCPs 2) Potential adverse health outcomes for the mother and child 3) Ways to reduce exposure

SUMMARY:
The purpose of this study is to reduce use of personal care products that contain endocrine disrupting chemicals among women. For this pilot intervention, the investigators focus on the hair care product class of personal care products, the reduction in use of phthalate-containing Hair Care Products (HCPs) and use among pregnant Women of Color (WOC).

DETAILED DESCRIPTION:
Endocrine disruptor chemicals (EDC) disrupt reproductive development and increase cancer risk through their ability to have a direct, indirect, or interactive action on cellular processes within the mammary tissues. EDCs may have the most influence during periods of dynamic structural and functional changes in the mammary glands, such as during pregnancy and the postpartum windows. Hair care products (HCPs) are a class of personal care products (PCPs) that contain EDCs; there are stark differences in HCP use by race. Differences in hair texture may explain differences in use. Nevertheless, of major concern, clinical, epidemiological, and laboratory studies have suggested HCPs are associated with earlier pubertal events, where the timing of pubertal maturation is an established risk factor for breast cancer (BC) risk. Additional studies have shown that compared to infrequent users, women classified as moderate or frequent users of PCPs had a 10-15% higher BC risk, dark hair dye is associated with a 52-72% increased BC risk, a history of chemical relaxer or straightener use is associated with a 64-74% increase in BC risk, and in 454 Mexican women (233 cases) urinary concentrations of monoethyl phthalate (MEP) were positively associated with BC, with stronger associations observed for pre-menopausal women. Evidence is emerging on EDC exposures across the pregnancy/postpartum periods. This is of importance because while pregnancy is associated with a long-term reduced risk of BC, it also confers an increased risk of BC for at least a decade after birth. EDC exposure during this period of increased risk could promote 'activation' effects for BC following pregnancy. In pregnant women, PCP use is correlated with higher concentrations of urinary phthalates, urinary metabolite concentrations vary by PCP type, and urinary metabolite concentrations differ by sociodemographic factors and across racial and ethnic populations.

Unfortunately, few studies examine HCP-associated EDC exposure across the pregnancy/postpartum periods and no study has implemented a behavioral intervention. An intervention during pregnancy on EDC exposures and HCPs could have intergenerational health implications.

An intervention to reduce phthalate exposures during the pregnancy/postpartum window would have both fetal/early and maternal health implications. First, behavioral changes during pregnancy could mitigate EDC exposures that exert in utero effects that may program long term risk for hormone-related disease for the child. Second, behavioral changes could reduce 'activation' effects for BC following pregnancy. Pregnant women are primed to change behaviors for their babies' health.

Therefore, the investigators propose an educational intervention for prenatal women of color in Northern Manhattan on HCPs and EDC exposures with an assessment of behavioral change via self-report and urinary phthalate concentrations.

ELIGIBILITY:
Inclusion Criteria:

* English and/or Spanish Speaking
* Pregnant women within first 4 weeks of 3rd trimester of pregnancy
* Lives within Northern Manhattan
* Women of color defined as Black or Hispanic women

Exclusion Criteria:

* Does not provide consent

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine A. McDonald, PhD, Principal Investigator — Columbia University
Locations (1):
- Community Engagement Core Community Space, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Yes: There is a plan to make individual participant data (IPD) and related data dictionaries available.
  Data and samples may be used by other Columbia researchers or researchers at other institutions for future research purposes. Participants name and other identifying information will have been permanently removed from the data and samples or the data and samples will be coded and the researchers who will use them will not have access to the key that links the code to the participant. Researchers who are not Columbia University Irving Medical Center (CUIMC) researchers on this study will only be given in de-identified or coded data.
Time Frame: End of study
Access Criteria: De-identified or coded data only.

REFERENCES:
- [Derived] Tsui F, Vilfranc CL, Llanos AAM, Houghton LC, Franklin J, More V, Manz KE, Pennell KD, Terry MB, Shepard P, Barrett E, Walker DAH, McDonald JA. Hair care product use among pregnant women of color: protocol for a feasibility educational intervention. Front Reprod Health. 2026 Jan 22;7:1694088. doi: 10.3389/frph.2025.1694088. eCollection 2025. PMID 41659359

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Educational Intervention
Started | 46
Completed | 31
Not Completed | 15
Not completed — Withdrawal by Subject | 15

BASELINE CHARACTERISTICS:
Groups:
- Educational Intervention Delivery and Change in Behavior: Educational Intervention: Deliver an educational intervention on harmful chemical exposures, such as phthalates, found in hair care products, developed by the research team using empirical evidence with key informant feedback. The intervention will cover phthalates 1) Exposure through HCPs 2) Potential adverse health outcomes for the mother and child 3) Ways to reduce exposure
Arm/Group | Educational Intervention Delivery and Change in Behavior
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 3
  More than one race | 17
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Change in Internal Dose of Urinary Phthalate Metabolites
Description: Urinary phthalate metabolites will be measured through gas chromatography-mass spectrometry (GC-MS). The percent change will be calculated from baseline to follow up 1 (FU1) and presented as a summary value of all low molecular weight phthalates (sumLMW). This outcome is calculated from the [(mean of FU1 - Mean of Baseline)/Mean of FU1]* 100. To calculate the sumLMW the investigators divided each metabolite by its molecular weight, summed the metabolites together, then multiplied by the average molecular weight of the metabolites.
Time Frame: Baseline (early Trimester 3 i.e. week 27-31 of pregnancy) and Follow up 1 (late Trimester 3 i.e. 4-6 weeks post baseline)
Population: 20 of 31 analyzed as urine samples were collected from 20 participants.
Measure: Mean (Standard Deviation); unit: percent change of sumLMW
Arm/Group | Educational Intervention
Number analyzed (Participants) | 20
percent change of sumLMW | 1.9 (0.7)

2. Primary Outcome: Change in Internal Dose of Urinary Phthalate Metabolites
Description: Urinary phthalate metabolites will be measured through gas chromatography-mass spectrometry (GC-MS). The percent change will be calculated from baseline to Follow up 2 (FU2) and presented as a summary value of all low molecular weight phthalates (sumLMW). This outcome is calculated from the [(mean of FU2 - Mean of Baseline)/Mean of FU2]* 100. To calculate the sumLMW the investigators divided each metabolite by its molecular weight, summed the metabolites together, then multiplied by the average molecular weight of the metabolites.
Time Frame: Baseline (early Trimester 3 i.e. week 27-31 of pregnancy) and Follow up 2 (1-month postpartum i.e. approx 3 months from baseline).
Population: 20 of 31 analyzed as urine sample were collected from 20 participants.
Measure: Mean (Standard Deviation); unit: percent change in sumLMW
Arm/Group | Educational Intervention Delivery and Change in Behavior
Number analyzed (Participants) | 20
percent change in sumLMW | -16.5 (1.3)

3. Secondary Outcome: Number of Participants With a Change in PAPM Stage
Description: Self reported behavioral changes as assessed by the Precaution Adoption Process Model (PAPM). The questionnaire allows investigators to assess the stage at each time point. The investigators will be examining PAPM as a change in stages: ΔPAPM (categorical). Label individual change by 1-stagnant (i.e. not moving from last reported stage); 2-regresses (i.e. regressing stage(s) from last reported stage) [cannot go back to unaware]; 3-progresses (i.e. advancing stage(s) from last reported stage; this will include Stage 4); 4th category will be included for a sub analysis if large enough, 4-negative-progresses. Category 3 is a best possible outcome and 2 is the worst possible outcome. The number of participants that show a change (progression) will be reported.
Time Frame: Baseline (early Trimester 3 i.e. week 27-31 of pregnancy ) and Immediate Post-Intervention (1-2 weeks post Baseline)
Population: 26 of 31 analyzed as 26 participants received the educational intervention and completed the baseline PAPM and the immediate post-PAPM.
Measure: Count of Participants; unit: Participants
Arm/Group | Educational Intervention
Number analyzed (Participants) | 26
Participants | 26

4. Secondary Outcome: Number of Participants With a Change in PAPM Stage
Description: as for outcome 3
Time Frame: Immediate Post-Intervention (1-2 weeks post Baseline) & Follow up 1 (late Trimester 3 i.e. 4-6 weeks post baseline)
Population: 12 of 31 analyzed as 12 participants completed the educational intervention and completed the immediate post intervention PAPM and the F/U1 PAPM
Measure: Count of Participants; unit: Participants
Arm/Group | Educational Intervention
Number analyzed (Participants) | 12
Participants | 9

5. Secondary Outcome: Number of Participants With a Change in PAPM Stage
Description: as for outcome 3
Time Frame: Follow up 1 (late Trimester 3 i.e. 4-6 weeks post baseline) & Follow-Up 2 (1-month postpartum i.e., approx 3 months from baseline)
Population: 7 of 31 analyzed as 7 participants completed the educational intervention and completed PAPM F/U1 and PAPM F/U2
Measure: Count of Participants; unit: Participants
Arm/Group | Educational Intervention
Number analyzed (Participants) | 7
Participants | 5

ADVERSE EVENTS:
Time Frame: Individuals were followed for adverse events over a maximum of 8 months.
Description: This is a minimum risk protocol.Participants will receive the following information about potential risks on the consent form: Participants may feel uncomfortable answering some of the questions on the questionnaires, but they have been informed that they have the right to refuse to respond to any questions they do not wish to answer.
Arm/Group | Educational Intervention
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT04493892/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT04493892/ICF_001.pdf